CLINICAL TRIAL: NCT01189994
Title: Pragmatic Randomized Controlled Trial of Acupuncture Effectiveness in the Treatment of Fibromyalgia
Brief Title: Trial of Acupuncture in the Treatment of Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Santa Casa da Misericordia do Rio de Janeiro Hospital (Other)
Responsible Party: Fernando Farias, MD, PhD, Santa Casa da Misericordia do Rio de Janeiro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCMRJH-001
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Fibromyalgia; Diffuse Myofascial Pain Syndrome; Fibromyalgia-Fibromyositis Syndrome; Fibromyositis-Fibromyalgia Syndrome; Myofascial Pain Syndrome, Diffuse
Keywords: Fibromyalgia; Acupuncture; Randomized Controlled Trial; Pain; Quality of Life
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Patients will receive acupuncture treatment in addition to standard care, coming to twelve weekly acupuncture sessions
  Interventions: Procedure: Acupuncture
- Orientation (Active Comparator): Patients will receive standard care only, coming to three monthly orientation sessions
  Interventions: Behavioral: Orientation

INTERVENTIONS:
Procedure: Acupuncture — Needling of acupoints, some of them receiving electrostimulation
  Arms: Acupuncture
Behavioral: Orientation — Orientation sessions focusing in fibromyalgia
  Arms: Orientation

SUMMARY:
Fibromyalgia is a medical condition characterized by musculoskeletal pain, fatigue, sleep disturbances and depression. It affects population at a socioeconomically active age and represents a burden for the patients and the health care system due to its personal and functional implications. At this moment, there is no completely effective treatment for fibromyalgia, and acupuncture has been a promising alternative. This trial aims to evaluate if addition of acupuncture to standard care represents an improvement in comparison with standard care only. Thus, patients enrolled in this trial will be randomly allocated into one of two groups: group A, who besides standard treatment will receive 12 sessions of acupuncture; and group B, who will receive standard care with monthly orientation sessions for the same period. Patients will be evaluated at baseline, after completion of acupuncture treatment or orientation, and after an additional 12-week follow up. Evaluation will be based on diaries of pain and medication, and standard scales of pain, quality of life and disability.

ELIGIBILITY:
Inclusion Criteria:

* American College of Rheumatology criteria for fibromyalgia
* elementary school
* drug treatment for at least 30 days (if any)

Exclusion Criteria:

* disabling mental condition
* other rheumatic conditions
* other chronic medical conditions with musculoskeletal symptoms
* pregnancy
* conditions that impair walking
* conditions that impair weekly consultations
* acupuncture treatment in the twelve-month period prior to enrollment
* diabetes mellitus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) score | Twelve weeks from baseline

SECONDARY OUTCOMES:
Weekly Likert scale in pain diary | Twelve weeks from baseline
Visual Analog Scale (VAS) for pain | Twelve weeks from baseline
Short Form 36 (SF-36) score for quality of life | Twelve weeks from baseline
Health Assessment Questionnaire - Disability Index (HAQ-DI) score | Twelve weeks from baseline
Hospital Anxiety and Depression (HAD) Scale | Twelve weeks from baseline
Fibromyalgia Impact Questionnaire (FIQ) score | Twenty-four weeks from baseline
Weekly Likert scale in pain diary | Twenty-four weeks from baseline
Visual Analog Scale (VAS) for pain | Twenty-four weeks from baseline
Short Form 36 (SF-36) score for quality of life | Twenty-four weeks from baseline
Health Assessment Questionnaire - Disability Index (HAQ-DI) score | Twenty-four weeks from baseline
Hospital Anxiety and Depression (HAD) Scale | Twenty-four weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Fernando P de Farias, MD, PhD, Principal Investigator — Santa Casa da Misericordia do Rio de Janeiro Hospital
Locations (1):
- Santa Casa da Misericordia do Rio de Janeiro Hospital; Instituto de Acupuntura do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil